CLINICAL TRIAL: NCT05925075
Title: Point of Care Lung Ultrasound in Preterm Infants with Respiratory Distress: a Multicenter Prospective Study
Brief Title: Point of Care Lung Ultrasound in Preterm Infants with Respiratory Distress
Status: Enrolling by invitation | Type: Observational
Sponsor: Phoenix Children's Hospital (Other)
Collaborators: MedStar Georgetown University Hospital (Other); Baylor Scott and White Health (Other); Children's Hospital Los Angeles (Other); St. Joseph's Hospital and Medical Center, Phoenix (Other); LAC+USC Medical Center (Other)
Responsible Party: Principal Investigator, Hemananda Muniraman, Staff Physician, Phoenix Children's Hospital
Other Study IDs: 22-176
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: lung ultrasound; BPD; bronchopulmonary dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- RDS: Infant born less than 32 weeks gestation with diagnosis of respiratory distress syndrome. Lung ultrasounds will be performed on day of life 7, 14, 21, 28 and at corrected gestational age of 36 weeks.
  Interventions: Diagnostic Test: Lung Ultrasound
- PDA: In addition to being less than 32 weeks gestation, subject can qualify for study and receive a lung ultrasound scan at time of echo diagnosis of patent ductus arteriosus (PDA).
  Interventions: Diagnostic Test: Lung Ultrasound
- Steroid: Aims are :
  A: To evaluate changes in LUS scores pre and post treatment with systemic steroid course.
  B: To evaluate the predictive ability of LUS for successful extubation following course of systemic steroids.
  Lung ultrasound scans will be done prior to initiation of post-natal steroid, day 1, day 3, day 7, day 10 of treatment and 1 week after steroid is discontinued.
  Interventions: Diagnostic Test: Lung Ultrasound

INTERVENTIONS:
Diagnostic Test: Lung Ultrasound — Lung ultrasound to be performed at scheduled intervals as described in individual cohorts.

SUMMARY:
The goal of this observational study is to learn about the role of bedside lung ultrasound in infants born prematurely with breathing problems. The main question this study aims to answer is: Can bedside lung ultrasound performed in the first month of life predict the development of chronic lung disease in premature infants?

DETAILED DESCRIPTION:
This is a multicenter study including preterm infants born less than 32 weeks gestational age and with a diagnosis of respiratory distress syndrome (RDS). Our primary aim is to determine the ability of lung ultrasounds performed in the first month of life to predict the development of bronchopulmonary dysplasia (BPD) at 36 weeks postmenstrual age.

Secondary aims will evaluate the association of lung ultrasound scores with the severity of hemodynamically significant patent ductus arteriosus (PDA) at time of diagnosis, as well as describe lung ultrasound changes pre and post-treatment with systemic steroid course.

Hypothesis:

1. LUS scores would have a predictive ability to identify extreme preterm infants at risk of BPD with AUC>0.8.
2. Higher LUS scores would correlate with higher severity of hemodynamically significant PDA.
3. LUS scores are expected to be lower after the course of systemic steroids and with lower scores are expected to predict successful extubation following the course of systemic steroids.

ELIGIBILITY:
Inclusion Criteria:

Infants born less than 32 weeks gestation and meet one or more of the below criteria A) Diagnosis of Respiratory Distress Syndrome B) Diagnosis of PDA C) Post-natal steroid treatment for the purpose of weaning off ventilation support

Exclusion Criteria:

Infants with critical congenital heart and lung conditions and those with genetic anomalies.

Min Age: 0 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All infants who are born less than 32 weeks gestation will be enrolled in the study after obtaining parent's consent.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Assess predictive ability of lung ultrasound scores in infants at risk of developing bronchopulmonary dysplasia (BPD) | The lung ultrasounds will be performed on day of life 7, 14, 21 and 28 and diagnosis of BPD would be per standard criteria.
  The primary outcome is to assess accuracy measures including specificity, sensitivity and area under ROC of lung ultrasound cut offs for predicting BPD.

SECONDARY OUTCOMES:
Association between lung ultrasound scores and severity of patent ductus arteriosus. | The lung ultrasound would be performed around the time of echocardiographic diagnosis of patent ductus arteriosus and severity determined by standard criteria.
  Secondary outcome is to assess correlation between lung ultrasound scores and severity of patent ductus arteriosus.
Comparison of lung ultrasound scores pre and post systemic steroid course administration | The lung ultrasound would be performed prior to steroid administration, 24 hours, 72 hours, 7 days, 10 days and 17 days after the first dose of 10 day course of systemic steroid administration.
  Comparison of lung ultrasound scores prior to and after course of systemic steroid administration would be analyzed using paired T-test or the signed Wilcoxon rank sum test.

CONTACTS AND LOCATIONS:
Locations (1):
- Phoenix Children's, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No